CLINICAL TRIAL: NCT03433079
Title: Incidence, Prediction and Time-dependent Role of Risk Factors of Acute Kidney Injury in Severe Trauma: Prospective Observational Cohort Study
Brief Title: Acute Kidney Injury in Severe Trauma
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-6
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Severe Trauma; NGAL; Tissue Hypoxia; Inflammatory Response; Rhabdomyolysis
MeSH Terms: conditions — Acute Kidney Injury; Wounds and Injuries; Rhabdomyolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Kidney Injury: Patients > 18 years of age with acute kidney injury were enroled into the study. Arterial levels of neutrophil gelatinase-associated lipocalin (NGAL), arterial lactate, interleukin-6 (IL-6), procalcitonin (PCT) and myoglobin were investigated in all patients.
  Interventions: Diagnostic Test: Neutrophil gelatinase-associated lipocalin (NGAL); Diagnostic Test: Arterial lactate; Diagnostic Test: Interleukin-6 (IL-6); Diagnostic Test: Procalcitonin (PCT); Diagnostic Test: Myoglobin

INTERVENTIONS:
Diagnostic Test: Neutrophil gelatinase-associated lipocalin (NGAL) — Blood neutrophil gelatinase-associated lipocalin (NGAL) test was performed in all patients.
Diagnostic Test: Arterial lactate — Arterial lactate level was assessed in all patients.
Diagnostic Test: Interleukin-6 (IL-6) — The level of interleukin-6 was assessed in all patients.
Diagnostic Test: Procalcitonin (PCT) — The level of procalcitonin (PCT) was assessed in all patients.
Diagnostic Test: Myoglobin — The level of myoglobin was assessed in all patients.

SUMMARY:
Acute kidney injury (AKI) represents a serious complication following severe injury associated with adverse outcome. Main goals of the presented study were to define the incidence of AKI and to evaluate the validity of AKI biomarker neutrophil gelatinase-associated lipocalin (NGAL) in AKI prediction in severely injured patients. Secondary goals were to determine the time-dependent role of injury-related tissue hypoxia, systemic inflammatory response, and rhabdomyolysis in the pathophysiology of AKI.

DETAILED DESCRIPTION:
The main goal of the presented study was to define the epidemiology of AKI and to evaluate the validity of AKI biomarker neutrophil gelatinase-associated lipocalin in AKI prediction in severely injured patients with Injury Severity Score (ISS) > 24. Secondary goals were to determine the time-dependent role of insults associated directly with the intensity of injury (tissue hypoxia, systemic inflammatory response and/or infection, rhabdomyolysis) in the pathophysiology of AKI.

The study was performed in a single center at the University Hospital in Ostrava in the Czech Republic. The Ethics Committee of the University Hospital Ostrava approved the study, which conformed to the tenets of the Declaration of Helsinki. Each of the awake and conscious study subjects signed the Informed Consent Form approved by the Ethics Committee of the University Hospital Ostrava. For enrolment of unconscious study subjects who were unable to sign informed consent, approval of two independent (i.e. not involved in the study) physicians was needed.

Patients and methods: All adult severely injured patients defined by Injury Severity Scale (ISS) > 24 admitted to the Department of Anaesthesiology and Intensive Care in University Hospital Ostrava between June 2013 and December 2015 were enrolled into the study. Subjects were screened for AKI presence defined by Kidney Disease: Improving Global Outcomes (KDIGO) criteria daily up to 8 days after injury. Arterial levels of neutrophil gelatinase-associated lipocalin (NGAL), lactate, interleukin-6 (IL-6), procalcitonin (PCT) and myoglobin were investigated at the time points 24 hours (T1), 48 hours (T2) and 96 hours (T3) after injury.

Methods All consecutive severely injured patients (ISS > 24) older than 18 years of age were enrolled in this prospective observational study between June 2013 and December 2015. All participants were admitted to the Level 1 Trauma Centre (Department of Anaesthesiology and Critical Care) at the University Hospital of Ostrava. Exclusion criteria included age < 18 years, history of kidney disease, pregnancy, death within 24 hours after injury, unsurvivable injury with an end of life decision (withhold or withdraw of therapy) pronounced within 24 hours after injury and, finally, clinical signs of brain death within 24 hours after injury.

Basic observed demographic parameters included age, ISS and mechanism of injury. The laboratory parameters included blood NGAL; arterial lactate level, IL-6, PCT and myoglobin at the 24 hours (T1), 48 hours (T2) and 96 hours (T3) after injury. Serum Creatinine level was assessed once daily at 6.00 a.m. and urine output collected hourly from admission (D0) to Day 8 were the basis for evaluation of AKI presence. Because of the recent pre-injury values of Creatinine were unknown almost in all of the subjects, first serum Creatinine level (sCr) taken on admission to the emergency room was used as a baseline reference value.

All diagnostic and therapeutic interventions were performed in accordance with guidelines and standards for the treatment of the critically injured patients. The study protocol does not contain any additional diagnostic or therapeutic intervention except the laboratory investigations mentioned above.

Early AKI defined according to KDIGO criteria occurs in one-third of victims of severe injury. Blood NGAL levels during the first 96 hours after injury are significantly higher in patients who subsequently develop AKI. Prolonged tissue hypoxia, excessive and prolonged activation of inflammatory response and rhabdomyolysis are factors contributing the development of AKI.

ELIGIBILITY:
Inclusion Criteria:

- severe injury (ISS >24)

Exclusion Criteria:

* age < 18 years
* history of kidney disease
* pregnancy
* death within 24 hours after injury
* unsurvivable injury (withheld or withdrawn therapy) within 24 hours after injury
* clinical signs of brain death within 24 hours after injury

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely injured patients (ISS > 24) older than 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury biomarker validity | 36 months
  The main goal of the study was to evaluate the validity of AKI biomarker neutrophil gelatinase-associated lipocalin in AKI prediction in severely injured patients with Injury Severity Score (ISS) > 24.

SECONDARY OUTCOMES:
Time-dependent role of insults | 36 months
  Secondary outcome measure was to determine the time-dependend role of insults associated directly with intensity of injury (tissue hypoxia, systemic inflammatory response and/or infection, rhabdomyolysis) in the pathopfysiology of AKI.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sklienka, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia